CLINICAL TRIAL: NCT01479946
Title: An International Randomized Phase II Study Comparing Early Electrochemotherapy to Delayed or No Electrochemotherapy in Patients With Cutaneous Breast Cancer Metastases
Brief Title: Electrochemotherapy For The Treatment Of Breast Cancer That Has Spread to the Skin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: ECT equipment not available at study center
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey Yachnin, Study Coordinator, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREATE-01
Record Dates: First submitted 2011-11-14; First posted 2011-11-28 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Skin Metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — Electrochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Electrochemotherapy (Experimental): Electrochemotherapy is given as early as possible after the discovery of skin metastases
  Interventions: Drug: Electrochemotherapy
- Delayed or no Electrochemotherapy (No Intervention): patients are to be treated for their breast cancer according to clinical routine with electrochemotherapy as an option only after 6 months from randomization

INTERVENTIONS:
Drug: Electrochemotherapy — bleomycin together with electroporation
  Arms: Early Electrochemotherapy

SUMMARY:
Electroporation combined with chemotherapy (ECT) has been shown to be an effective treatment for breast cancer that has spread to skin. In routine clinical practise, ECT is offered to patients when all other treatment options have been exhausted. This study tests the hypothesis that early treatment with ECT may result in improved local control of skin metastases, improved quality of life and reduced health care costs. Patients are randomised to either ECT given as early as possible in the course of the disease or delaying ECT for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age
* Histological confirmed breast cancer
* Metastatic breast cancer (skin lesions only are considered as metastatic disease)
* Prior histological confirmation of at least one skin lesion
* Skin lesions must not have a depth greater than 3 cm (measured clinically if possible otherwise on the basis of CT/ultrasound examination
* Confluent skin metastases where individual lesions are hard to define in their entirety may not exceed a maximum area of 10 x 10 cm for each area of confluence. If there are several areas of confluence, the patient may be included in the study provided that all lesions can be treated within the time constraints of a single ECT session (20 minutes).
* Not more than ten skin lesions. Each area of confluence is considered as one lesion.
* A single skin lesion may not exceed 5 cm
* Patients may not have received more than one line of systemic treatment (chemotherapy or endocrine therapy) for metastatic disease following the discovery of skin metastases. Patients developing skin metastases for the first time during ongoing systemic therapy may receive one additional line of systemic treatment prior to inclusion.
* Patients in the early ECT arm may receive any other cancer treatments at the discretion of the treating physician starting no earlier than 2 weeks following ECT. This is to ensure that patients with metastatic disease in other locations will receive treatment that is considered suitable regardless of their participation in this trial. (If 2 weeks from ECT to the start of systemic treatment is judged to be too long by the treating physician, this patient should not be entered into the trial).
* Women of childbearing age must practice a suitable form of contraception.
* A life expectancy of at least 6 months.
* Patients with a ECOG performance status < 3
* Signed Informed Consent

Exclusion Criteria:

* Patients who have extensive and rapidly progressive visceral metastases where a delay in systemic therapy by eventual ECT is judged to not be in the patients' best interest
* Patients, who for medical reasons, cannot be given bleomycin
* Patients with brain metastases treated with surgery and/or radiotherapy who have progressive disease in the brain two months after treatment
* Prior cumulative dose of bleomycin exceeding 250,000 IU/m2
* Less than 14 days from previous cancer treatment (either local or systemic)
* If the patient has skin lesions that are situated in close proximity to a pacemaker such that an electrical field from ECT will overlap the pacemaker, the pacemaker must be moved to another location in order for the patient to be able to participate in the study
* Chronic renal failure (serum creatinine > 150 mol/L)
* Inadequate liver function defined as:

ASAT or ALAT > 2.5 x ULN in the absence of liver metastases or > 5 in the presence of liver metastases or Bilirubin > 2 x ULN (except in the case of Gilberts Syndrome) or Albumin < 25 g/L

• Inadequate bone marrow reserve defined as: White blood cell count < 3 X 109/L or Neutrophil count < 1.5 X109/L or Platelet count < 100 X 109/L

* Any severe uncontrolled systemic disease.
* Unable or unwilling to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
local control of skin metastases | 6 months from randomisation

SECONDARY OUTCOMES:
Local control of skin metastases during the time interval of 6 to 18 months after randomization | 18 months
  The same measurement for local control as the primary endpoint
Quality of Life | monthly (up to 18 months)
  EQ5D and FACT-B questionaires are to be filled on a monthly basis throughout the 18 month study period
Health economic analysis | recorded monthly (up to 18 months)
  the number of out-patient visits, duration of hospital admissions if any, the number of type of systemic therapies, frequency of medical imaging and when applicable, the requirement for sick-leave.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Yachnin, MD, PhD, Study Director — Uppsala University Hospital
Locations (1):
- Deaprtment of Oncology, University Hospital Uppsala, Uppsala, Sweden